CLINICAL TRIAL: NCT05717452
Title: Effects of a Single Dose of Wild Blueberries on Mood and Executive Function in Healthy Emerging Adults: a Single-Blind, Randomized Controlled Trial
Brief Title: Effects of a Single Dose of Wild Blueberries on Mood and Executive Function in Healthy Emerging Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Prof. Claire Williams, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-140-RC
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mood; Affect; Executive Function
Keywords: Blueberry; Anthocyanins

STUDY DESIGN:
Intervention Model Description: Standard two-arm trial with a placebo arm and active intervention arm
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry drink (Experimental)
  Interventions: Dietary Supplement: Blueberry drink
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Blueberry drink — 22 g freeze-dried wild blueberry (Vaccinium angustifolium) powder mixed with 250 ml water.
  Arms: Blueberry drink
Dietary Supplement: Placebo drink — 22 g placebo powder matched for macronutrients, color, and flavor mixed with 250 ml water.
  Arms: Placebo drink

SUMMARY:
This study aims to investigate whether consuming a drink containing powdered blueberries (equivalent to 150 g of fresh fruit) can improve mood and executive function in healthy emerging adults.

DETAILED DESCRIPTION:
The present study will examine the psychological effects of a single dose of freeze-dried wild blueberries using a randomized, single-blind, placebo-controlled design. A total of 80 participants will be randomly allocated to consume either a drink prepared with 22 g blueberry powder or a drink prepared with 22 g placebo powder matched for macronutrients, flavour and colour.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years of age

Exclusion Criteria:

* Any medically significant condition or mental health disorder (e.g. diabetes, endocrine or gastrointestinal disorders)
* Taking medication (excluding hormonal contraception or medication for asthma/seasonal allergies)
* Allergy to blueberries or any other Vaccinium species

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Positive affect as measured by PANAS-X | 1.5 hours post-ingestion
  Positive affect will be calculated by adding the values of the 21 positive items of the Positive and Negative Affect Schedule-X and the additional item "motivated". Thus, the scale will range from 0 to 88 points with higher scores indicating better mood.

SECONDARY OUTCOMES:
Negative affect as measured by PANAS-X | 1.5 hours post-ingestion
  Negative affect will be calculated by adding the values of the 25 negative items of the Positive and Negative Affect Schedule-X. Thus, the scale will range from 0 to 100 points with higher scores indicating worse mood.
Executive function (accuracy) | 1.5 hours post-ingestion
  A task-switching test will be used to assess cognitive flexibility when switching between two predictable tasks requiring simple numerical decisions. The main outcome of interest is the average accuracy (0 to 100%).
Reaction time | 1.5 hours post-ingestion
  The average reaction time on correct trials of the task-switching test (in milliseconds).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT05717452/Prot_SAP_000.pdf